CLINICAL TRIAL: NCT05661409
Title: The Use of Sugammadex as Rescue Therapy Following Inadequate Reversal With Neostigmine
Brief Title: Sugammadex as Rescue Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Georgia Clinical & Translational Science Alliance (CTSA) (Unknown)
Responsible Party: Principal Investigator, Matthew K Whalin, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004369; UL1TR002378 (NIH)
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Neuromuscular Blockade
Keywords: Neostigmine; Sugammandex
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Sugammadex 2 mg/kg (Active Comparator): The study team will identify patients who are scheduled to undergo an elective surgery under general anesthesia, received rocuronium for NMB and neostigmine for NMB reversal.
  Patients will be randomized using the Emory University REDCap (Research Electronic Data Capture) software to six groups: 2 mg/kg (the lowest dose approved by the FDA), 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg, 0.125 mg/kg of sugammadex and placebo. Doses would be based on actual body weight. The time taken to reach a TOF ratio of 0.9 thereafter would be measured. If the patient fails to achieve this goal by 10 minutes, sugammadex would be given in 2 mg/kg increments until the patient reaches this threshold and can be safely extubated. The TOF ratio would be measured again at 30 minutes after arrival at the PACU to exclude delayed residual NMB with the plan to give further 2 mg/kg doses of sugammadex if detected.
  Interventions: Drug: Sugammadex
- Sugammadex 1 mg/kg (Experimental): The study team will identify patients who are scheduled to undergo an elective surgery under general anesthesia, received rocuronium for NMB and neostigmine for NMB reversal.
  Patients will be randomized using the Emory University REDCap (Research Electronic Data Capture) software to six groups: 2 mg/kg (the lowest dose approved by the FDA), 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg, 0.125 mg/kg of sugammadex and placebo. Doses would be based on actual body weight. The time taken to reach a TOF ratio of 0.9 thereafter would be measured. If the patient fails to achieve this goal by 10 minutes, sugammadex would be given in 2 mg/kg increments until the patient reaches this threshold and can be safely extubated. The TOF ratio would be measured again at 30 minutes after arrival at the PACU to exclude delayed residual NMB with the plan to give further 2 mg/kg doses of sugammadex if detected.
  Interventions: Drug: Sugammadex
- Sugammadex 0.5 mg/kg (Experimental): The study team will identify patients who are scheduled to undergo an elective surgery under general anesthesia, received rocuronium for NMB and neostigmine for NMB reversal.
  Patients will be randomized using the Emory University REDCap (Research Electronic Data Capture) software to six groups: 2 mg/kg (the lowest dose approved by the FDA), 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg, 0.125 mg/kg of sugammadex and placebo. Doses would be based on actual body weight. The time taken to reach a TOF ratio of 0.9 thereafter would be measured. If the patient fails to achieve this goal by 10 minutes, sugammadex would be given in 2 mg/kg increments until the patient reaches this threshold and can be safely extubated. The TOF ratio would be measured again at 30 minutes after arrival at the PACU to exclude delayed residual NMB with the plan to give further 2 mg/kg doses of sugammadex if detected.
  Interventions: Drug: Sugammadex
- Sugammadex 0.25 mg/kg (Experimental): The study team will identify patients who are scheduled to undergo an elective surgery under general anesthesia, received rocuronium for NMB and neostigmine for NMB reversal.
  Patients will be randomized using the Emory University REDCap (Research Electronic Data Capture) software to six groups: 2 mg/kg (the lowest dose approved by the FDA), 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg, 0.125 mg/kg of sugammadex and placebo. Doses would be based on actual body weight. The time taken to reach a TOF ratio of 0.9 thereafter would be measured. If the patient fails to achieve this goal by 10 minutes, sugammadex would be given in 2 mg/kg increments until the patient reaches this threshold and can be safely extubated. The TOF ratio would be measured again at 30 minutes after arrival at the PACU to exclude delayed residual NMB with the plan to give further 2 mg/kg doses of sugammadex if detected.
  Interventions: Drug: Sugammadex
- Sugammadex 0.125 mg/kg (Experimental): The study team will identify patients who are scheduled to undergo an elective surgery under general anesthesia, received rocuronium for NMB and neostigmine for NMB reversal.
  Patients will be randomized using the Emory University REDCap (Research Electronic Data Capture) software to six groups: 2 mg/kg (the lowest dose approved by the FDA), 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg, 0.125 mg/kg of sugammadex and placebo. Doses would be based on actual body weight. The time taken to reach a TOF ratio of 0.9 thereafter would be measured. If the patient fails to achieve this goal by 10 minutes, sugammadex would be given in 2 mg/kg increments until the patient reaches this threshold and can be safely extubated. The TOF ratio would be measured again at 30 minutes after arrival at the PACU to exclude delayed residual NMB with the plan to give further 2 mg/kg doses of sugammadex if detected.
  Interventions: Drug: Sugammadex
- Placebo (Placebo Comparator): The inclusion of a placebo group would allow the study team to examine if patients may recover spontaneously over that time without needing any sugammadex at all, and what parameters may predict that subset of patients. It will also improve the dose response modelling, in that randomization has been weighted so that patients who are least likely to need sugammadex (i.e. if they achieved a TOF count of 4 twitches without fade) are more likely to be in the placebo group or at the lowest dose of sugammadex that is being tested.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sugammadex — Sugammadex is a FDA-approved drug that is in routine clinical use for NMB reversal.
  Patients will be randomized to six groups: 2 mg/kg (the lowest dose approved by the FDA), 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg, 0.125 mg/kg of sugammadex and placebo. Doses would be based on actual body weight. The time taken to reach a TOF ratio of 0.9 thereafter would be measured. If the patient fails to achieve this goal by 10 minutes, sugammadex would be given in 2 mg/kg increments until the patient reaches this threshold and can be safely extubated.
  Arms: Sugammadex 0.125 mg/kg; Sugammadex 0.25 mg/kg; Sugammadex 0.5 mg/kg; Sugammadex 1 mg/kg; Sugammadex 2 mg/kg
Drug: Placebo — Normal saline will be used as placebo. The inclusion of a placebo group would allow us to examine if patients may recover spontaneously over that time without needing any sugammadex at all, and what parameters may predict that subset of patients. It will also improve the dose response modelling, in that randomization has been weighted so that patients who are least likely to need sugammadex (i.e. if they achieved a TOF count of 4 twitches without fade) are more likely to be in the placebo group or at the lowest dose of sugammadex that is being tested.
  Arms: Placebo

SUMMARY:
Neuromuscular blocking agents (NMBAs) are commonly used in the practice of anesthesiology for skeletal muscle relaxation to facilitate tracheal intubation, mechanical ventilation, and to provide optimal surgical conditions. In order to prevent residual NMB, it is vital to adequately reverse any use of a non-depolarizing NMBA. This was historically done using an anticholinesterase such as neostigmine, which would increase the concentration of acetylcholine at the neuromuscular junction leading to the return of neuromuscular transmission. Unfortunately, there are disadvantages to the use of an anticholinesterase. It was in this context that sugammadex was found to be a valuable addition to the anesthesiologist's armamentarium. It is a modified γ-cyclodextrin that encapsulates the aminosteroid NMBAs rocuronium and vecuronium.

This project is a double-blind randomized placebo-controlled dose-response trial that aims to determine the time taken to achieve adequate reversal comparing five doses of sugammadex as rescue therapy following inadequate reversal with neostigmine. The study team will recruit patients aged 18 years and above from the main operating room and outpatient surgery center at Grady Memorial Hospital who are undergoing elective surgery under general anesthesia, who has received NMB, received neostigmine for NMB reversal, and achieved a TOF count ≥ 3 twitches but not a TOF ratio of 0.9 fifteen minutes after neostigmine was given. Those with a TOF count < 3 twitches will drop out of the study as there are already specified doses of sugammadex for that level of NMB

DETAILED DESCRIPTION:
Neuromuscular blocking (NMB) agents are commonly used in the practice of anesthesiology for skeletal muscle relaxation to facilitate tracheal intubation, and may require reversal in order to prevent residual NMB. This was historically done using an anticholinesterase such as neostigmine, which has many adverse effects and may not effectively reverse a deep NMB. However, the introduction of sugammadex was instrumental in allowing the rapid return of neuromuscular function. The FDA has only approved three doses of sugammadex (2 mg/kg, 4 mg/kg and 16 mg/kg) depending on the train of four (TOF) count, which is a qualitative measure of the depth of NMB and ranges from 0 to 4 twitches. Conversely, the TOF ratio is a quantitative measure, is calculated using the ratio of the amplitude of the fourth twitch to the first twitch, and ranges from 0 to 1. A TOF ratio of 0.9 is generally accepted as the minimum threshold to safely extubate a patient, but this information is not always readily accessible as many anesthesia providers do not have a quantitative NMB monitor.

In 2020, Carvalho et al. conducted a meta-analysis of 53 studies (12,664 adult patients) where the pooled residual NMB incidence ranged from 0.115 when quantitative neuromuscular monitoring was used to 0.331 where no neuromuscular monitoring was used. Ravel et al. conducted a meta-analysis of 20 randomized controlled trials (1,923 adult patients), where residual NMB was found in 2.8% of patients who received sugammadex compared to 39% of those who received neostigmine 15 minutes post administration. Concerningly, 60 minutes after administration, 2.1% of the sugammadex group versus 19% of the neostigmine group still had NMB. When expanded to observational studies (58 studies with 25,277 adult patients), the incidence of residual NMB ranged from 0% to 90.5% (median 30%), which was significantly lower (0% to 16%) in the sugammadex group compared to 3.5% to 90.5% in the neostigmine group and 15% to 89% in the spontaneous recovery group.

This project is a double-blind randomized placebo-controlled dose-response trial that aims to determine the time taken to achieve adequate reversal comparing five doses of sugammadex as rescue therapy following inadequate reversal with neostigmine. The study team will recruit patients aged 18 years and above from the main operating room and outpatient surgery center at Grady Memorial Hospital who are undergoing elective surgery under general anesthesia, who has received NMB, received neostigmine for NMB reversal, and achieved a TOF count ≥ 3 twitches but not a TOF ratio of 0.9 fifteen minutes after neostigmine was given. Those with a TOF count < 3 twitches will drop out of the study as there are already specified doses of sugammadex for that level of NMB.

These patients will then be randomized to six groups: 2 mg/kg (the lowest dose approved by the FDA), 1 mg/kg, 0.5 mg/kg, 0.25 mg/kg, 0.125 mg/kg of sugammadex, and placebo. The time taken to reach a TOF ratio of 0.9 thereafter would be measured and compared for statistically significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above who will undergo an elective surgery in the main operating room or outpatient surgery center at Grady Memorial Hospital
* Receive general anesthesia (standardized to sevoflurane for maintenance)
* Receive rocuronium for NMB
* Receive neostigmine for NMB reversal
* Achieve a TOF count of at least 3 twitches but not a TOF ratio of 0.9 fifteen minutes after neostigmine has been given
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy and/or lactating
* BMI ≥ 40
* Severe renal impairment, i.e. chronic kidney disease stages IV and V as defined by GFR < 30 ml/min/1.73 m2
* Severe hepatic impairment, i.e. Child-Pugh score C
* Pre-existing neuromuscular disease
* Anticipated need for postoperative intubation, and/or known hypersensitivity reactions to rocuronium, neostigmine and/or sugammadex.
* Adults unable to consent
* Prisoners
* Cognitively impaired or Individuals with Impaired Decision-Making Capacity
* Individuals who are not able to clearly understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Whalin, MD, Principal Investigator — Assistant Professor
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.
  Proposals should be directed to Dr. Whalin at mwhalin@emory.edu To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Grady Memorial Hospital OR who were scheduled to undergo an elective surgery under general anesthesia, received rocuronium for NMB, and received neostigmine for NMB reversal, and achieved a TOF count of at least 3 twitches but had a TOF ratio less than 0.9 15 minutes after neostigmine had been given. Participant enrollment began on July 21, 2023, and the final study assessment occurred on August 2, 2024.
Groups:
- Sugammadex 2 mg/kg; Sugammadex 1 mg/kg; Sugammadex 0.5 mg/kg; Sugammadex 0.25 mg/kg; Sugammadex 0.125 mg/kg; Placebo: Patients were randomized to one of the six dose-based groups. The groups were differentiated based on dose given per kg of body weight
Period: Overall Study
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 1 mg/kg | Sugammadex 0.5 mg/kg | Sugammadex 0.25 mg/kg | Sugammadex 0.125 mg/kg | Placebo
Started | 8 | 7 | 6 | 7 | 8 | 10
Completed | 7 | 6 | 6 | 6 | 6 | 6
Not Completed | 1 | 1 | 0 | 1 | 2 | 4
Not completed — Drug administered, but monitor disconnected | 1 | 0 | 0 | 0 | 0 | 0
Not completed — No TOFR data; problem with the monitor | 0 | 1 | 0 | 0 | 0 | 0
Not completed — TOFR≥0.9 at time of drug admin. | 0 | 0 | 0 | 1 | 2 | 2
Not completed — Lost TOFR data prior to time study drug given | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Miscommu-nication about administration | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 1 mg/kg | Sugammadex 0.5 mg/kg | Sugammadex 0.25 mg/kg | Sugammadex 0.125 mg/kg | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 6 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (15.9) | 58.8 (17.2) | 52.0 (13.9) | 50.2 (10.2) | 56.7 (14.1) | 44.8 (15.8) | 53.0 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 3 | 3 | 5 | 4 | 23
  Male | 4 | 1 | 3 | 3 | 1 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 5 | 6 | 6 | 5 | 34
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 5 | 5 | 4 | 6 | 6 | 33
  White | 0 | 1 | 0 | 2 | 0 | 0 | 3
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
BMI [Count of Participants; unit: Participants]
  <20 kg/m^2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  20-29 kg/m^2 | 5 | 2 | 4 | 3 | 2 | 4 | 20
  30-39 kg/m^2 | 2 | 4 | 2 | 3 | 3 | 2 | 16
ASA Status [Count of Participants; unit: Participants] — The ASA status is assigned by the anesthesiologist on the day of surgery, after assessing the patient's medical history, physical examination, and other relevant factors.
  ASA I: A normal, healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life
  Participants
    ASA I | 1 | 0 | 0 | 0 | 0 | 0 | 1
    ASA II | 0 | 1 | 3 | 0 | 2 | 3 | 9
    ASA III | 6 | 5 | 3 | 6 | 4 | 3 | 27
    ASA IV | 0 | 0 | 0 | 0 | 0 | 0 | 0
Surgery duration [Mean (Standard Deviation); unit: minutes] | 261 (81) | 260 (96) | 303 (103) | 239 (70) | 209 (74) | 207 (77) | 247 (85)
Total rocuronium [Mean (Standard Deviation); unit: mg] | 111 (46) | 84 (44) | 130 (56) | 113 (24) | 77 (27) | 82 (28) | 100 (42)
Neostigmine dose [Mean (Standard Deviation); unit: mg/kg] | 4.57 (0.53) | 4.08 (1.43) | 4.25 (0.99) | 4.50 (0.84) | 4.58 (0.80) | 4.08 (1.11) | 4.35 (0.93)
Time from last rocuronium to neostigmine [Mean (Standard Deviation); unit: mins] | 53.1 (29.5) | 59.0 (44.3) | 48.5 (18.0) | 63.7 (24.6) | 81.3 (19.8) | 58.5 (51.5) | 60.5 (32.8)
Baseline train-of-four ratio TOFR (0-1) [Mean (Standard Deviation); unit: units on a scale] — The ratio of the fourth response T4 to the first response T1. Range is 0 to 1. Best outcome is 1, indicating no residual neuromuscular block
  units on a scale | 1.00 (0) | 1.00 (0) | 1.00 (0) | 1.00 (0) | 1.00 (0) | 0.99 (0.02) | 1.00 (0.01)
Train-of-four count (TOFC) before neostigmine [Count of Participants; unit: Participants] — The number of twitches as detected by the anesthesia provider. Range is 0 twitch, 1 twitch, 2 twitches, 3 twitches, 4 twitches with fade, 4 twitches without fade. Best outcome is 4 twitches without fade, suggesting no residual neuromuscular block
  Participants
    0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    1 | 2 | 1 | 1 | 2 | 2 | 1 | 9
    2 | 1 | 1 | 2 | 1 | 3 | 1 | 9
    3 | 2 | 0 | 0 | 0 | 0 | 2 | 4
    4 with fade | 2 | 3 | 3 | 2 | 1 | 2 | 13
    4 without fade | 0 | 1 | 0 | 1 | 0 | 0 | 2
Train-of-four ratio (TOFR) before neostigmine (0-1) [Mean (Standard Deviation); unit: units on a scale] — The ratio of the fourth response T4 to the first response T1. Range is 0 to 1. Best outcome is 1, indicating no residual neuromuscular block
  units on a scale | 0.04 (0.12) | 0.00 (0.00) | 0.06 (0.09) | 0.00 (0.00) | 0.04 (0.09) | 0.02 (0.06) | 0.03 (0.08)
Train-of-four count (TOFC) 15 mins after neostigmine [Count of Participants; unit: Participants] — Range is 0 twitch, 1 twitch, 2 twitches, 3 twitches, 4 twitches with fade, 4 twitches without fade. Best outcome is 4 twitches without fade, suggesting no residual neuromuscular block.
  Participants
    0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    4 with fade | 1 | 0 | 0 | 0 | 2 | 2 | 5
    4 without fade | 6 | 6 | 6 | 6 | 4 | 4 | 32
Train-of-four ratio (TOFR) before study drug (0-1) [Mean (Standard Deviation); unit: units on a scale] — The ratio of the fourth response T4 to the first response T1. Range is 0 to 1. Best outcome is 1, indicating no residual neuromuscular block.
  units on a scale | 0.47 (0.31) | 0.57 (0.14) | 0.65 (0.10) | 0.52 (0.32) | 0.65 (0.14) | 0.69 (0.21) | 0.59 (0.22)
Train-of-four ratio (TOFR) 15 mins after neostigmine (0-1) [Mean (Standard Deviation); unit: units on a scale] — The ratio of the fourth response T4 to the first response T1. Range is 0 to 1. Best outcome is 1, indicating no residual neuromuscular block.
  units on a scale | 0.48 (0.30) | 0.55 (0.14) | 0.64 (0.12) | 0.52 (0.32) | 0.58 (0.21) | 0.63 (0.20) | 0.56 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: The Time Taken to Achieve a TOF Ratio of 0.9 After Administration Sugammadex
Description: The time taken to achieve a time of train (TOF) ratio of 0.9 after the use of the intervention drug versus placebo in a patient population that has already received neostigmine for NMB reversal.
  Quantitative neuromuscular monitoring will be carried out using electromyography, which measures the TOF ratio every 20 seconds. The TOF count (between 0 to 4) and the TOF ratio (0 to 1) would be measured and recorded at baseline and after administration of the study drug. If the TOF ratio remains < 0.9 after this, or if the patient exhibits any symptoms or signs of residual NMB blockade, a further 2 mg/kg dose of sugammadex would be given until the patient achieves a TOF ratio of 0.9.
Time Frame: 10 minutes post administration of study drug
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 1 mg/kg | Sugammadex 0.5 mg/kg | Sugammadex 0.25 mg/kg | Sugammadex 0.125 mg/kg | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 6
minutes | 3.13 (3.15) | 2.56 (0.96) | 2.33 (0.84) | 5.00 (3.97) | 4.94 (2.64) | 9.67 (0.82)

2. Secondary Outcome: The Percentage of Patients Who Achieve a TOF Ratio of 0.9
Description: The percentage of patients who achieve a TOF ratio of 0.9 will be measured within 1 minute, 2 minutes, 5 minutes, and 10 minutes after the administration of the study drug, sugammadex.
Time Frame: 1 minute, 2 minutes and 10 minutes post administration of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 1 mg/kg | Sugammadex 0.5 mg/kg | Sugammadex 0.25 mg/kg | Sugammadex 0.125 mg/kg | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 6
Participants
  in 1 min | 2 | 1 | 1 | 1 | 0 | 0
  in 2 min | 4 | 2 | 2 | 2 | 0 | 0
  in 5 min | 6 | 6 | 6 | 4 | 5 | 1
  in 10 min | 7 | 6 | 6 | 4 | 5 | 1

ADVERSE EVENTS:
Time Frame: The time frame is up to the time the patient is transferred out of the PACU. This occurs when an anesthesiologist determines that the patient has recovered from anesthesia and typical durations are 1-2 hours.
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 1 mg/kg | Sugammadex 0.5 mg/kg | Sugammadex 0.25 mg/kg | Sugammadex 0.125 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6 | 2/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/7 | 3/6 | 0/6 | 3/6 | 2/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugammadex 2 mg/kg (N=7) | Sugammadex 1 mg/kg (N=6) | Sugammadex 0.5 mg/kg (N=6) | Sugammadex 0.25 mg/kg (N=6) | Sugammadex 0.125 mg/kg (N=6) | Placebo (N=6)
Hypotension (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugammadex 2 mg/kg (N=7) | Sugammadex 1 mg/kg (N=6) | Sugammadex 0.5 mg/kg (N=6) | Sugammadex 0.25 mg/kg (N=6) | Sugammadex 0.125 mg/kg (N=6) | Placebo (N=6)
Nausea (General disorders) | 0 | 3 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT05661409/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT05661409/ICF_000.pdf